CLINICAL TRIAL: NCT07260682
Title: Effect of Probiotic Supplementation on Renal Function, Vascular Calcification and Alterations in Bone Mineral Metabolism in Patients With Chronic Kidney Disease
Acronym: MICKID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PI20/0660; PI20/0660 (Other Grant/Funding Number: ISCIII)
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease (Stages 3b-5)
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Probiotic — Supplement: Lactobacillus DMG0017 Probimel Dosage: 15 ml/day for 6 months. Directions: Take alone or diluted in juice, any sugary drink, or yogurt. Pharmaceutical Form: Lactobacillus oral solution Route of administration: oral

SUMMARY:
INTRODUCTION You have been asked to participate in a research study of patients with chronic kidney disease to assess whether a probiotic supplement (a commercially available product that is not a medication) can help slow the progression of your vascular calcification and thus improve your health. Your participation in this study does not replace your usual medical care.

Why is this study being conducted? The purpose of this study is to demonstrate that a probiotic supplement is helpful in slowing the progression of your vascular calcification. We also intend to assess whether changes in vascular calcification are associated with changes in mineral metabolism parameters, inflammation, and kidney function.

What does the study involve? This study will include patients with chronic kidney disease and vascular calcification.

Half of the patients will receive the probiotic supplement Probimel at a dose of 15 ml per day. The study will last 6 months, during which time your kidney function, vascular calcification, and parameters related to uremic toxins, inflammation, and mineral metabolism will be evaluated. The study physician may adjust the dosage of your usual medication before you begin using the study food product, or during the study if your symptoms change. Please ask your study physician or team any questions you may have.

STUDY PROCEDURES If you agree to participate in this study and sign this Consent Form, you will undergo some tests during a screening period to determine if you are eligible to participate. This screening takes place before your inclusion in the main phase of the study.

At each study visit, you will be asked about:

* any medications you are currently taking or any changes to them,
* any problems you are experiencing,
* any side effects you may be having, which may or may not be related to the study,
* whether you have visited any other doctors or hospitals.

Following the explanation of the research project and the signing of informed consent during the initial screening visit, the patient's medical history will be reviewed, anthropometric measurements will be taken, and existing biochemical data will be analyzed.

During the first visit, blood will be drawn, stool samples will be collected, and the degree of vascular calcification will be assessed using abdominal, pelvic, and hand X-rays. The study and treatment with the probiotic supplement will begin at this point.

Subsequent visits will be scheduled at 2 and 6 months, during which blood samples (hematology and biochemistry) will be taken. Additionally, at the final visit (month 6), stool collection and X-rays will be repeated.

At this point, treatment will be discontinued, and the study will be concluded, with a final follow-up visit scheduled to ensure that all studied parameters are stable and within the normal range. Excess blood samples from this study will be stored in the Biobank of the Reina Sofía University Hospital in Córdoba and may be used later in other scientific studies. For this reason, you will receive an additional document in which you give your consent for the proper storage of the samples in the biobank.

What should I do during the study?

To obtain reliable information from this study on the effect of probiotic supplementation in patients with chronic kidney disease and vascular calcification, you are expected to do the following:

* Follow your study physician's instructions.
* Attend all scheduled study visits and complete all procedures.
* Review all medications you are taking with your study physician. Certain medications you are currently taking or have taken in the past may prevent you from participating in this study.
* Some procedures/illnesses you have had in the past may prevent you from participating in this study. • Take and store your study medication as directed, and return any leftover medication and/or empty containers to your doctor at each visit.
* Do not share your study medication with anyone. You are the only person authorized to take it.
* Keep your study medication and materials out of the reach and sight of children and anyone who cannot read or understand all the information about it.
* Tell the study staff about any health problems you have, even if you think they are not important.
* Tell the study staff if you wish to stop participating in this study.
* Do not participate in any other research studies.

ELIGIBILITY:
Inclusion Criteria:

1. Be of legal age (≥18 years).
2. Patients with stage 5 CKD in pre-dialysis or dialysis with evidence of cardiovascular disease. Calcification will be quantified using the Kaupilla and Adragao indices as indicated in Appendix 1. All radiographs necessary to assess the degree of calcification (both at the beginning and end of the study) will be examined by the same radiologist. To avoid bias in the assessments, the calculation of the Adragao and Kaupilla indices will be performed by staff from the Radiology Department of the Reina Sofía University Hospital.
3. Negative pregnancy test.
4. Patient capable of understanding the study procedures and who provides informed consent to participate in the research project.

Exclusion Criteria:

1 Patients diagnosed with or suspected of having inflammatory bowel disease.

2. Patients undergoing antibiotic treatment within the last two months prior to the start of the study.

3. Patients with recurrent infections or diverticula treated intermittently with antibiotics.

4. No cardiovascular history.

5. Other cardiovascular or metabolic disorders.

6. Pregnant or breastfeeding women, or women planning to become pregnant.

7. Drug or alcohol addiction that, in the investigator's opinion, could interfere with compliance with the study requirements.

8. Participation in other clinical studies.

9. Incapacity or unwillingness of the individual, legal guardian, or representative to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
To analyze the effect of probiotic supplementation | 6 months
  To analyze the effect of probiotic supplementation on the progression of vascular calcification during chronic kidney disease

CONTACTS AND LOCATIONS:
Locations (1):
- IMIBIC, Córdoba, Andalusia, Spain